CLINICAL TRIAL: NCT04621864
Title: Can Gene Polymorphisms Influence Morphine Analgesic Consumption After Laparoscopic Cholecystectomy? A Prospective Cohort Study.
Brief Title: Gene Polymorphisms and Morphine Analgesic Consumption
Status: Completed | Type: Observational
Sponsor: Hamad Medical Corporation (Industry)
Collaborators: Qatar University (Other)
Responsible Party: Sponsor
Other Study IDs: MRC-01-18-270
Record Dates: First submitted 2020-08-07; First posted 2020-11-09 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2021-11

CONDITIONS: Gene; Polymorphosis
Keywords: Gene; Polymorphisms;morphine;analgesia;laparoscopic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Withdraw a 5 ml blood sample just after induction anesthesia. This sample will be stored at the refrigerator at 4 °C till handled to one of our research coordinator at faculty of pharmacy at QU.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Variation of morphine requirements are seen considerably. Studies showed that pharmacogenetics (PGx) could possibly be used to tailor pain medication according to an individual's genetic background. While prior studies demonstrated the association of genetic polymorphism with opioid requirements in various types of surgeries in Asian and European populations, there are no published data in Middle East populations especially Arabs. However, in our area we have a lot of theincity that may give us an answer for this research question.

Objectives: The primary Objective of this study is to investigate whether the genetic polymorphism of human μ-opioid receptor gene (OPRM1), ATP binding cassette gene (ABCB1) and rs2952768 are contributing to the variation of morphine consumption in women undergoing laparoscopic cholecystectomy. The secondary objective is to assess the effect of these genetic polymorphisms on pain score, analgesic dosage requirements, and complications of morphine use in these patients within the first 24 hours.

DETAILED DESCRIPTION:
Background: Variation of morphine requirements are seen considerably. Studies showed that pharmacogenetics (PGx) could possibly be used to tailor pain medication according to an individual's genetic background. While prior studies demonstrated the association of genetic polymorphism with opioid requirements in various types of surgeries in Asian and European populations, there are no published data in Middle East populations especially Arabs.

Objectives: The primary Objective of this study is to investigate whether the genetic polymorphism of human μ-opioid receptor gene (OPRM1), ATP binding cassette gene (ABCB1) and rs2952768 are contributing to the variation of morphine consumption in women undergoing laparoscopic cholecystectomy. The secondary objective is to assess the effect of these genetic polymorphisms on pain score, analgesic dosage requirements, and complications of morphine use in these patients within the first 24 hours.

Methods: This is a pilot prospective cohort study to be conducted at Al-Wakrah Hospital, HMC after receiving IRB approval from MRC. The aim is to recruit 100 adult female Arab patients with American Society of Anesthesiologists physical status of I or II in whom planned postoperative pain management by morphine will be requested after laparoscopic cholecyctectomy Baseline demographic information will be collected at baseline along with 4ml blood sample for genotyping. Morphine will be administered repeatedly for postoperative pain relief and the total dose administered within the first 24 hours will be collected. The analgesic effect will be evaluated using a visual analogue scale (VAS). Multiple linear regression will be used to evaluate the association of the genetic variant groups with the morphine dose and the pain score after adjusting for different confounders. Logistic regression will be used to evaluate the association of side effect of vomiting and respiratory depression with the genetic variants. Baseline characteristic values will be reported as mean ± SD for continuous variables or frequency and percentage for categorical variables. A priori P value of ≤ 0.05 will be considered significant. All analyses will be done using the Statistical version 25 of SPSS software.

ELIGIBILITY:
Inclusion Criteria:

* . They agree to participate and sign the informed consent

  * They are older than 18 years
  * They are women undergoing laparoscopic cholecystectomy.

Exclusion Criteria:

* . They have significant respiratory, cardiovascular, renal, hepatic diseases or diabetes.

  * They have history of allergy to morphine and those with bad experience to morphine side effects.
  * They have chronic pain and those taking pain medications.

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — To rule out Gender factor in pain
Study Population: After the approval of the our institutional review board committee IRB at HAMAD MEDICAL CORPORATION (HMC), Doha, Qatar, and written, informed consent, 100 adult female patients with American Society of Anesthesiologists physical status of I or II in whom planned postoperative pain management by morphine will be requested after laparoscopic cholecystectomy can will be included in this study; at the Wakrah Hospital, HMC. We planned to study 300 patients. If a genetic abnormality was found in 15% of patients and the average total morphine use in this subgroup was 40% lower than in the remainder of the patients, then there was 80% chance that a t test comparing average log-total morphine would be significant at P ≤ 0.05.
Sampling Method: Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2020-11-20 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
genetic polymorphism of human Opioid receptors | Day One (D1)
  The primary Objective of this study is to investigate whether the genetic polymorphism of human μ-opioid receptor gene (OPRM1), ATP binding cassette gene (ABCB1) and rs2952768 are contributing to the variation of morphine consumption in women undergoing laparoscopic cholecystectomy.

SECONDARY OUTCOMES:
The effect of genetic polymorphisms on pain score and analgesic dosage requirements | Day One (D1)
  The secondary objective is to assess the effect of these genetic polymorphisms on pain score, analgesic dosage requirements, and complications of morphine use in these patients within the first 24 hours.

CONTACTS AND LOCATIONS:
Overall Officials: HAMED ELGENDY, MD,PhD, Principal Investigator — Consultant Anesthesia - HMC & Associate Prof Anesthesia - Qatar University - Adjunct A-Prof Weill Conel Medicine Qatar
Locations (1):
- HAMAD Medical Corporation- Al Wakra Hospital, Doha, Select, Qatar

REFERENCES:
- [Derived] Elgendy HM, Ibrahim SM, Bader L, Mohammad RA, Ali ZO, Bejaoui MBA, Hilani M, Ismail H, Elewa HF. Genetic Factors Associated with Morphine Consumption in Women Undergoing Laparoscopic Cholecystectomy: A Prospective Cohort Study. J Pain Res. 2023 Jul 15;16:2407-2417. doi: 10.2147/JPR.S420447. eCollection 2023. PMID 37456358